CLINICAL TRIAL: NCT04277832
Title: Evaluation of a New Screening Tool (TUPAST) for Psoriatic Arthritis in Turkish Psoriasis Population and Comparison With TOPAS 2 for Validation of TUPAST
Brief Title: Evaluating of New Screening Tool for Arthritis* in Psoriasis
Acronym: TUPAST
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 54022451-050.05.05
Record Dates: First submitted 2020-02-03; First posted 2020-02-20 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Psoriasis; Psoriatic Arthritis
Keywords: psoriasis; psoriatic arthritis; screening tool
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single arm: Group of psoriasis patients will select randomly. All selected psoriasis patients will be consulted to a physician experienced in rheumatology and all of patients will fill TUPAST and TOPAS 2 forms.
  Interventions: Diagnostic Test: Questionary

INTERVENTIONS:
Diagnostic Test: Questionary — All patients will answer two different questionary (TUPAST, TOPAS 2)

SUMMARY:
This study evaluates a new screening tool for arthritis in psoriasis and compares its reliability with well-known screening tool (TOPAS 2).

DETAILED DESCRIPTION:
Early diagnosis and treatment of PsA may prevent destruction in joints.Our aim is to create a simple and user friendly screening tool that can be used by dermatologists in out patient clinics.

A question pool will be created from a review of the literature and expert opinions from a physicians experienced in rheumatology and dermatologists .Psoriasis patients will answer these newly created questions. All patients will be examined by dermatology and also physical therapy and rehabilitation-rheumatology experts. The diagnosis of psoriatic arthritis (PsA) will be made by CASPAR (Classification criteria for psoriatic arthritis) criteria and ASAS (Assessment of Spondyloarthritis International Society) criteria for spondyloarthritis. Synchronously patients will be asked for to reply Turkish version of well known questionary named TOPAS 2. According to the results of collected data, statistically best matched questions will be selected for Turkish population. Also, the reliability of TUPAST (Turkish PsA Screening Tool) and TOPAS 2 (Toronto Psoriatic Arthritis Screen II) will be compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis confirmed by dermatologist

Exclusion Criteria:

* Unable to consent and understand
* Known other rheumatological disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years with psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Creation of new tool (TUPAST: Turkish psoriatic arthritis screening tool) for detecting psoriatic arthritis among psoriasis patients | six months, throughout the study
  Questions which related with psoriatic arthritis will be selected statistically. Factor analysis will be performed to select the questions to construct the questionnaire. ROC (receiver operating characteristic) will be used to pick the best cut point for tool. Then, sensitivity and specificity of new tool to detect psoriatic arthritis among psoriasis patients will be calculated.
Correlation between TOPAS 2 score and probability of psoriatic arthritis in psoriasis patients | six months, throughout the study
  TOPAS 2 (Toronto Psoriatic Arthritis Screen II ) is a questionnaire for detecting psoriatic arthritis which has 95.8% sensitivity and 98% specificity in Turkish population. All patients will answer TOPAS 2 questions and all patients will be examined by dermatology and also physical therapy and rehabilitation-rheumatology experts.The diagnosis of psoriatic arthritis (PsA) will be made by CASPAR (Classification criteria for psoriatic arthritis) criteria and ASAS (Assessment of Spondyloarthritis International Society) criteria for spondyloarthritis.Then, sensitivity and specificity of TOPAS 2 will be calculated in our group and the correlation between psoriatic arthritis and screening tool results will be seen.
Comparison of the reliability of the TUPAST and TOPAS 2 | six months, throughout the study
  All patients will answer TUPAST and TOPAS 2 at the same time. According to statistical results, reliability of this two tool will be compared.
Correlation between TUPAST score and probability of psoriatic arthritis in psoriasis patients | six months, throughout the study
  All patients will answer TUPAST questions and all patients will be examined by dermatology and also physical therapy and rehabilitation-rheumatology experts.The diagnosis of psoriatic arthritis (PsA) will be made by CASPAR (Classification criteria for psoriatic arthritis) criteria and ASAS (Assessment of Spondyloarthritis International Society) criteria for spondyloarthritis. Then, sensitivity and specificity of TOPAS 2 will be calculated in our group and the correlation between psoriatic arthritis and screening tool results will be seen.

SECONDARY OUTCOMES:
Demographic characteristics demographic characteristics demographic characteristics | six months
  Demographic characteristics of patients will be compared (especially between PsA and non PsA group)

CONTACTS AND LOCATIONS:
Overall Officials: Nahide MD Onsun, Prof, Study Director — Bezmialem University; Begüm MD Güneş, Principal Investigator — Bezmialem University
Locations (1):
- Bezmialem Vakıf Univesity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Husni ME, Meyer KH, Cohen DS, Mody E, Qureshi AA. The PASE questionnaire: pilot-testing a psoriatic arthritis screening and evaluation tool. J Am Acad Dermatol. 2007 Oct;57(4):581-7. doi: 10.1016/j.jaad.2007.04.001. Epub 2007 Jul 3. PMID 17610990
- [Background] Ibrahim GH, Buch MH, Lawson C, Waxman R, Helliwell PS. Evaluation of an existing screening tool for psoriatic arthritis in people with psoriasis and the development of a new instrument: the Psoriasis Epidemiology Screening Tool (PEST) questionnaire. Clin Exp Rheumatol. 2009 May-Jun;27(3):469-74. PMID 19604440
- [Background] Chiowchanwisawakit P, Wattanamongkolsil L, Srinonprasert V, Petcharat C, Siriwanarangsun P, Katchamart W. Developing the Thai Siriraj Psoriatic Arthritis Screening Tool and validating the Thai Psoriasis Epidemiology Screening Tool and the Early Arthritis for Psoriatic Patients questionnaire. Rheumatol Int. 2016 Oct;36(10):1459-68. doi: 10.1007/s00296-016-3513-4. Epub 2016 Jun 22. PMID 27333800
- [Background] Audureau E, Roux F, Lons Danic D, Bagot M, Cantagrel A, Dernis E, Gouyette N, Hilliquin P, Jullien D, Liote F, Passeron T, A Richard M, Claudepierre P. Psoriatic arthritis screening by the dermatologist: development and first validation of the 'PURE-4 scale'. J Eur Acad Dermatol Venereol. 2018 Nov;32(11):1950-1953. doi: 10.1111/jdv.14861. Epub 2018 Mar 9. PMID 29430720
- [Result] Duruoz MT, Sanal Toprak C, Ulutatar F. Validation of the Toronto Psoriatic Arthritis Screen II (TOPAS II) questionnaire in a Turkish population. Rheumatol Int. 2018 Feb;38(2):255-259. doi: 10.1007/s00296-017-3871-6. Epub 2017 Nov 7. PMID 29116441